CLINICAL TRIAL: NCT02795026
Title: To Investigate the Use of Trans-perineal Trigger Point Dry Needling With Manual Therapy and to Compare the Outcome With Manual Therapy Treatment for Chronic Pelvic Pain With Dyspareunia. A Randomized Clinical Trial.
Brief Title: Trans-perineal Trigger Point Dry Needling for Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cork University Hospital (Other)
Collaborators: University College Cork (Other)
Responsible Party: Principal Investigator, Shalini Wiseman, Senior Physiotherapist in Women's Health & Continence, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115224510
Record Dates: First submitted 2016-06-04; First posted 2016-06-09 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Dyspareunia
Keywords: dry needling; vulvodynia; pelvic pain chronic
MeSH Terms: conditions — Dyspareunia; Vulvodynia | interventions — Musculoskeletal Manipulations; Myofascial Release Therapy

STUDY DESIGN:
Masking Description: It is difficult to mask the participants or care provider due to the nature of the therapy. The outcome questionnaires are filled in individually by the participants only.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual therapy (Active Comparator): Intervention to be administered is manual therapy with myofascial release of trigger points for pelvic floor muscles, pelvis and abdominal musculature.
  Interventions: Procedure: Manual therapy
- Dry needling & manual therapy (Active Comparator): Intervention to be administered is Trans-perineal trigger point dry needling, done externally to target the trigger points in the pelvic floor muscles along with dry needling of the pelvis and abdominal musculature.Manual therapy will only be used in areas difficult to reach with the acupuncture needles.
  Interventions: Procedure: Manual therapy; Procedure: Trigger point dry needling

INTERVENTIONS:
Procedure: Manual therapy — Myofascial trigger point release technique is a technique used to help ease tight muscles. This technique involves palpating the tight muscle for the 'knot'/trigger point and gently applying pressure for 30-60 seconds to help ease out the trigger point.
  Other Names: myofascial release
Procedure: Trigger point dry needling — Trigger point dry needling is a treatment technique involving the use of a single, disposable, fine filament acupuncture needle. Here the tight muscle is palpated and the acupuncture needle is directed towards the trigger point. The insertion of the needle is not felt, however the twitch reflex elicited to ease off the trigger point can be felt . This can be sore, but lasts only for a few seconds. Trans-perineal trigger point dry needling is an effective dry needling technique for the pelvic floor muscles done externally, targeting the trigger points in the pelvic floor muscles.
  Other Names: intra-muscular therapy; deep dry needling; trans-perineal trigger point dry needling
  Arms: Dry needling & manual therapy

SUMMARY:
Chronic Pelvic Pain (CPP) are around 10% of gynaecology referrals.Non-relaxing pelvic floor dysfunction (NRPFD) is an under-appreciated cause for CPP with dyspareunia where no other pathology exists. The effectiveness of manual therapy in studies have shown statistically significant pre and post treatment differences.However no study has reviewed the efficacy of inclusion of trans- perineal trigger point dry needling used with manual therapy for NRPFD. This study will investigate the effectiveness of trans-perineal trigger point dry needling used with manual therapy techniques for CPP.

DETAILED DESCRIPTION:
This study will investigate the effectiveness of inclusion of trans-perineal trigger point dry needling with manual therapy treatment for chronic pelvic pain with dyspareunia and associated pelvic floor dysfunctions.The use of trigger point dry needling (TrptDN) for chronic low back pain has proved beneficial.This study will evaluate the treatment outcomes of trans-perineal trigger point dry needling and manual therapy to only manual therapy for CPP.

The outcomes will evaluate the number of treatment requirements between the dry needling with manual therapy group and the manual therapy group and review which group has faster resolution in pain and other associated pelvic floor symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients reporting non-cyclical CPP with dyspareunia and associated PFD with no palpable pelvic floor pathology, but with palpable high pelvic floor muscle (PFM) tone and tenderness will be referred for physiotherapy by the gynaecology team.
* Visceral conditions like interstitial cystitis are difficult to exclude at gynaecology review, as they mimic CPP symptoms.
* Smokers and non-smokers included.
* Nulliparous, singleton and multiparous patients.

Exclusion Criteria:

* Body mass index greater than 30, makes it difficult to dry needle as the required needle length is not available.
* Chronic back pain over 6 months duration, under pain management team.
* Orthopaedic back surgeries with implants.
* Pelvic pathologies like endometriosis, fibroids, cysts, etc.
* Pregnancy related pelvic pain.
* Pregnant during the trial.
* Pelvic organ carcinomas.
* Undergoing cancer treatment.
* Post gynaecology surgeries, less than 16 weeks.
* Cardiovascular, gastroenterology, renal or orthopaedic surgery, less than 6 month's post-operative.
* Neurological conditions like stroke, epilepsy, Parkinson's disease etc.
* Exclusion criteria for dry needling:
* Extreme needle phobia, Rheumatoid arthritis, prolonged corticosteroid treatment, warfarin treatment, heart implants and blood clotting disorders.
* Participant with no significant learning disability and should be able to understand the procedure to consent for treatment.
* Participant should not require a chaperone during treatment.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2016-04; Primary Completion 2018-04-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Pain reduction or resolution within 10 treatment sessions, evaluated with the 0-10 Numeric Pain Rating Scale (0-10NPRS) | 10 weeks or earlier on resolution
  Participants will be asked to fill the 0-10NPRS at base line, 4th, 8th and 10th session or earlier on resolution of symptoms and to review which arm has faster resolution with lesser treatment sessions.

SECONDARY OUTCOMES:
Resolution in dyspareunia | 10 weeks or earlier on resolution
  Evaluated with the Female Sexual Functional Index questionnaire (FSFI) at baseline and the 10th session or earlier on resolution
Resolution in bladder, bowel and sexual dysfunction | 10 weeks or earlier on resolution
  Evaluated with the abbreviated International Pelvic Pain Questionnaire (IPPQ) concentrating on dyspareunia and painful bladder and bowel symptoms. This is done at baseline and at 10th session or earlier as per resolution.
Patient treatment satisfaction in each group | 10 weeks or earlier on resolution
  Evaluated with Pain Treatment Satisfaction Scale (PTSS) at 10th session or earlier on resolution

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne O'Sullivan, Dr., Principal Investigator — Cork University Maternity Hospital; Louise Kenny, Prof, Principal Investigator — Cork University Maternity Hospital
Locations (2):
- Ireland (2):
  - Cork University Maternity Hospital, Cork, Co.Cork
  - Cork Womens Clinic, Cork, Co.Cork

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT02795026/Prot_SAP_000.pdf